CLINICAL TRIAL: NCT06146686
Title: Clinical Effectiveness of Single Rotary File Versus Multiple Rotary Files in Pulpectomy of Primary Molars : A Randomized Clinical Trial
Brief Title: Single Rotary File Pulpectomy in Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Eid Ahmed Elsayed, doctor , internal resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: single rotary file pulpectomy
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Pulpitis - Irreversible
Keywords: single rotary file pulpectomy , primary molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The blinding of the operator is not possible due to the nature of the technique used. Trial participants, outcome assessors and statistician will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I ( pulpectomy using single rotary file ) (Experimental): After opening the access cavity, a single rotary file (20 taper 4) will be adjusted on the desirable working length depending on a radiograph (1 mm shorter than the apex) and used in pulpectomy in a brushing motion at the rotational speed 300 rpm with torque set at the lowest level, irrigation with saline
  Interventions: Device: Fanta AF blue rotary files 20 taper 4
- Group II ( pulpectomy using multiple rotary files system ) (Active Comparator): After opening the access cavity, multiple rotary files system (Fanta AF baby rotary files 20 taper 4, 25 taper 4, 30 taper 4) will be adjusted on the desirable working length depending on a radiograph (1 mm shorter than the apex) and used in pulpectomy in a brushing motion at rotational speed 300 rpm with torque set at the lowest level, irrigation with saline
  Interventions: Device: Fanta AF baby rotary files 20 , 25 , 30 taper 4

INTERVENTIONS:
Device: Fanta AF blue rotary files 20 taper 4 — single rotary file Fanta AF blue rotary files 20 taper 4
  Arms: Group I ( pulpectomy using single rotary file )
Device: Fanta AF baby rotary files 20 , 25 , 30 taper 4 — multiple rotary files system Fanta AF baby rotary files 20 , 25 , 30 taper 4
  Arms: Group II ( pulpectomy using multiple rotary files system )

SUMMARY:
The aim of this study is to compare the clinical effectiveness of a single rotary file system versus a multiple rotary files system in pulpectomy of primary molars

DETAILED DESCRIPTION:
In pediatric dentistry, premature loss of necrotic primary molars has been a matter of great concern over the years.

In modern pedodontic practice, Pulpectomy is regarded as the choice modality of treatment for pulpally involved necrotic teeth.

Hand files are used for mechanical preparation of primary tooth during pulpectomy but it has been found to be time consuming and may negatively influence the child's behavior . Much attention has been directed toward making pulpectomy a less time-consuming and a more-efficient procedure.

These challenges lead to the introduction of rotary endodontics in pediatric dentistry. However, the bizarre root canal morphology and thinner root dentin limited the use of rotary endodontics in primary teeth. Various modified protocols have been introduced to overcome such barriers to prevent undesirable complications.

Up to our knowledge, no clinical trials in the literature have been done to compare the clinical and radiographic success of single rotary file systems versus multiple rotary files systems when used in pulpectomy of primary molars. Thus, the present study aims to investigate the clinical effectiveness of those two techniques

ELIGIBILITY:
Inclusion Criteria:

* Children Criteria:

  * Medically free .
  * Cooperative patient.

Molar criteria :

• Mandibular second primary molar with clinical signs or symptoms of irreversible pulpitis

Radiographic criteria:

* No evidence of internal/external pathologic root resorption.
* With or without periapical or furcal lesion .

Exclusion Criteria:

* • Uncooperative children.

  * Children with systemic disease.
  * Lack of informed consent by the child patient's parent.
  * Refusal of participation.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
instrumentation time | during the operation
  instrumentation time of pulpectomy using single rotary file by stopwatch

SECONDARY OUTCOMES:
child's cooperation level | baseline and during the operation
  child's cooperation level using Frenkel's behaviour rating scale using Grades ( 1- Definitely negative 2- negative 3- positive 4- definitely positive )
obturation quality | immediately after the operation
  obturation quality measuring using periapical radiographs using Coll and Sadrian criteria ( scores) the quality of the root canal filling was defined as :
  1. underfilling : all the canals were filled more than 2 mm short of the apex
  2. optimal filling : one or more of the canals having the obturant ending at the radiographic apex or up to 2 mm short of the apex
  3. overfilling : any canal showing obturant outside the root

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Kohli A, Chhabra J, Sharma K, Katyayan R, Bhatnagar P, Sharma A. Comparative Evaluation of Instrumentation Time and Quality of Obturation amongst Pediatric Rotary Endodontic System: An In Vivo Study. Int J Clin Pediatr Dent. 2023 Mar-Apr;16(2):338-343. doi: 10.5005/jp-journals-10005-2573. PMID 37519962
- [Background] Kalita S, Agarwal N, Jabin Z, Anand A. Comparative Evaluation of Cleaning Capacity and Efficiency of Kedo-S Pediatric Rotary Files, Rotary ProTaper, and Hand K Files in Primary Molar Pulpectomy. Int J Clin Pediatr Dent. 2021 May-Jun;14(3):383-387. doi: 10.5005/jp-journals-10005-1958. PMID 34720511